CLINICAL TRIAL: NCT00257023
Title: Exploratory Study of Paliperidone in Patients With Schizophrenia to Investigate the Safety and Efficacy
Brief Title: An Exploratory Study on the Safety and Effectiveness of Paliperidone in Patients With Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR004939
Record Dates: First submitted 2005-11-18; First posted 2005-11-22 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2011-01

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Risperidone; Positive and Negative Syndrome Scale (PANSS); Clinical Global Impression (CGI); Positron Emission Tomography (PET)
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate

INTERVENTIONS:
Drug: paliperidone

SUMMARY:
The purpose of this study is to assess the safety, effectiveness, and plasma concentration of paliperidone (an antipsychotic medication) given once daily in the treatment of patients with schizophrenia

DETAILED DESCRIPTION:
Paliperidone is an extended-release tablet. Paliperidone is an active metabolite of risperidone, not approved for the treatment of schizophrenia in Japan. This is a multicenter, open-label, parallel-group, fixed dose study to evaluate the safety, effectiveness, and plasma concentration of paliperidone taken once daily in patients with schizophrenia. The patients will receive a fixed dose of paliperidone (3, 9, and 15 mg) for 6 weeks and its effectiveness and safety will be observed for an additional 2 weeks.. Efficacy will be measured by determining changes throughout the study in the Positive and Negative Syndrome Scale (PANSS) score, a scale for the measurement of symptoms of schizophrenia, and the Clinical Global Impression (CGI) score. In addition, the study also assesses the relationship between dose/plasma drug concentration and dopamine D2 receptor occupancy in patients who consent to receive positron emission tomography (PET). Safety evaluations (symptoms, physical exams, electrocardiograms, laboratory tests, Drug-Induced Extrapyramidal Symptoms Scale [DIESS] results, and adverse event monitoring) will be conducted throughout the study. The study hypothesis is that paliperidone will be effective in the treatment of schizophrenia, and that it will be well-tolerated. The patients will receive either 3, 9, or 15 mg of paliperidone, taken once daily by mouth for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with schizophrenia according to the diagnostic criteria of DSM-IV
* taking not more than one oral antipsychotic medication within 28 days of study entry
* a score below 120 at pre-treatment on the Positive and Negative Syndrome Scale Score (PANSS), a scale for the measurement of symptoms of schizophrenia

Exclusion Criteria:

* Diagnosis of psychiatric disease other than schizophrenia according to the diagnostic criteria of DSM-IV
* history of Parkinson's disease, seizure disorder, cerebrovascular accident, diabetes mellitus, clinically significant gastrointestinal disorders, or severe impairment of the liver or kidneys
* drug allergy or hypersensitivity to antipsychotics

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2005-02; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Safety assessments conducted throughout the study, including adverse events and results from the Drug-Induced Extrapyramidal Symptoms Scale [DIESS]

SECONDARY OUTCOMES:
Changes measured throughout the study in the Positive and Negative Syndrome Scale (PANSS) score, a score on a scale for the measurement of symptoms of schizophrenia, and the Clinical Global Impression (CGI) score.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K. Clinical Trial, Study Director — Janssen Pharmaceutical K.K.

REFERENCES:
- See also: Exploratory study of JNS007ER in patients with Schizophrenia to investigate the Safety and Efficacy. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=408&filename=CR004939_CSR.pdf